CLINICAL TRIAL: NCT05462925
Title: Point-of-care Prediction of Muscle Responsiveness to Functional Electrical Stimulation Therapy During Neurorehabilitation (sub-study)
Brief Title: Prediction of Muscle Responsiveness to FES Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Wings for Life (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-5395
Record Dates: First submitted 2022-07-04; First posted 2022-07-18 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Spinal cord injury; Functional electrical stimulation; Upper limb; Electromyography; Prediction.
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This prognostic study examines how baseline measurements predict therapy response in a single group of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Functional electrical stimulation therapy (Experimental): Participants will receive 30 sessions of upper limb functional electrical stimulation therapy. Sessions will be 1 hour in length and take place 3-5 times per week.
  Interventions: Device: Functional electrical stimulation therapy.

INTERVENTIONS:
Device: Functional electrical stimulation therapy. — Functional electrical stimulation therapy will be delivered using the MyndMove system (MyndTec, Inc., Mississauga, Canada).

SUMMARY:
Reduced arm and hand function has a significant impact on independence and quality of life after spinal cord injury. Functional electrical stimulation therapy (FES-T) is a treatment that can produce improvements in reaching and grasping function after neurological injuries. However, not all paralyzed muscles respond equally well to the therapy. Currently, therapists cannot predict which muscles will respond, limiting their ability to create a personalized therapy plan that can maximize outcomes while making the best use of the limited treatment time available. The objective of this study is to develop a diagnostic method that will allow therapists to quickly and easily screen muscles in the clinic, in order to predict how they will respond to FES-T.

Participants with cervical spinal cord injury will receive FES-T through the Rocket Family Upper Extremity Clinic at the Toronto Rehabilitation Institute - University Health Network. Muscles receiving training will undergo a electrophysiological examination before the start of therapy, and will then be tracked for strength recovery over the course of 30 sessions. Lastly, signal processing and machine learning techniques will be applied to the electrophysiological data to predict the recovery profile of each muscle.

The significance of this work will be to provide personalized therapy planning in FES-T, leading to more effective use of healthcare resource as well as improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Cervical spinal cord injury
* Paralysis or paresis in at least one upper extremity
* At least 6 months post SCI
* Able to understand and follow instructions
* Able to tolerate being in a seated position for a least one hour required to deliver upper limb therapy
* Willing to attend treatment sessions and all assessment sessions
* Able to understand and provide informed consent
* Male and female participants ≥ 18 years of age at the time of enrollment

Exclusion Criteria:

* Previous history of any other neuromuscular disorder or conditions that may affect motor response
* Upper extremity injury or condition prior to SCI that limits the function of the hand or arm
* In the judgment of the medical provider, the participant has medical complications that may interfere with the execution of the study
* Currently enrolled in another upper limb study and/ or has received MyndMove Therapy within the past 3 months
* Botulinum toxin injection into affected upper extremity and the muscle targeted by MyndMove® therapy within 3 months prior to the study start. No botulinum toxin injections in the upper extremity during the study treatment.
* Females who are pregnant or planning to become pregnant in the duration of the trial
* Regional disorder of the upper extremities such as fracture, dislocation, or joint contractures to less than 50% of the expected range of motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle strength recovery profile | Muscle strength assessed at each of 30 therapy sessions (3-5 sessions per week).
  Change over time in manual muscle testing conducted on each treated muscle.

SECONDARY OUTCOMES:
Surface electromyography signal features | Baseline (required). End of therapy (6-10 weeks; optional).
  Surface electromyography of treated muscles will be conducted at baseline. A set of signal features will be extracted for use in predictive modeling (examples include Hudgins' time-domain feature set, autoregressive coefficients, and frequency domain features). An optional second assessment will occur at the end of the 30 therapy sessions.

CONTACTS AND LOCATIONS:
Overall Officials: José Zariffa, PhD, Principal Investigator — University Health Network, Toronto; Sukhvinder Kalsi-Ryan, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared following study completion upon reasonable request to the investigators and completion of a data sharing agreement.
Time Frame: Once study has been published, the datasets corresponding to the analyses described will be shared upon request.
Access Criteria: Data sharing will require completion of a data sharing agreement. Interested parties should contact the principal investigator.

REFERENCES:
- [Derived] Balbinot G, Li G, Chen A, Eftekhar P, Ma W, Kalsi-Ryan S, Zariffa J. Upper Extremity Muscle Recovery Profiles With Functional Electrical Stimulation Therapy in Chronic Spinal Cord Injury. Neuromodulation. 2025 Oct 16:S1094-7159(25)01026-8. doi: 10.1016/j.neurom.2025.08.416. Online ahead of print. PMID 41099684